CLINICAL TRIAL: NCT00151762
Title: A Multi-Center, 52-Week, Open-Label Extension Study (From Studies WEL-301, WEL-302, and WEL-303) to Evaluate the Long-Term Safety and Tolerability of WelChol® in Type 2 Diabetic Patients
Brief Title: Long-Term Study of Safety and Efficacy of WelChol® as an Additional Therapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Kenneth Truitt, Daiichi Sankyo
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: WEL-304
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Type 2 Diabetes
Keywords: Open label, Diabetes Mellitus; Long term safety study, extension study
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Colesevelam hydrochloride

SUMMARY:
This extension study is designed to evaluate the long-term safety and tolerability of colesevelam hydrochloride (WelChol®) in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion/Rollover Criteria:

* Patients who have completed studies WEL-301, WEL-302, or WEL-303 with treatment compliance at least 80%
* Patients who have completed studies WEL-301, WEL-302, or WEL-303 who have not met withdrawal criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of colesevelam hydrochloride as add-on therapy

SECONDARY OUTCOMES:
To assess the long-term effect on hemoglobin A1c
To assess the long-term effect on fasting plasma glucose
To assess effects on lipids and lipoproteins

CONTACTS AND LOCATIONS:
Locations (64):
- United States (62):
  - Birmingham, Alabama
  - Tuscumbia, Alabama
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Carmichael, California
  - Concord, California
  - Irvine, California
  - La Jolla, California
  - Los Angeles, California
  - Los Gatos, California
  - San Diego, California
  - Spring Valley, California
  - West Hills, California
  - Washington D.C., District of Columbia
  - Cocoa Beach, Florida
  - Coral Gables, Florida
  - Largo, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Troy, Michigan
  - Edina, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Bozeman, Montana
  - Butte, Montana
  - Las Vegas, Nevada
  - Rochester, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Marion, Ohio
  - Perrysburg, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Bristol, Tennessee
  - Morristown, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Lakewood, Washington
- Mexico City, Mexico
- Lima, Peru